CLINICAL TRIAL: NCT07101042
Title: A Comparative Study of Cold and Paraspinal Stimulation on Erectile Dysfunction and Urinary Incontinence in Spinal Cord Injury Patients
Brief Title: Cold vs. Paraspinal Stimulation for Erectile and Urinary Function in SCI Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Hassan Fayed, Physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Erectile Dysfunction; Urinary Incontinence; Paraspinal Stimulation; Cold Therapy;
MeSH Terms: conditions — Spinal Cord Injuries; Erectile Dysfunction; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups. The first group received localized cold stimulation, while the second group received paraspinal electrical stimulation. Both interventions were applied independently, with no crossover between groups throughout the study period.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor was blinded to group allocation. Participants and care providers were aware of the intervention being delivered due to the physical nature of the treatments (cold vs. electrical stimulation). The blinded assessor was responsible for administering and scoring all post-treatment outcome measures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Stimulation (Experimental): Participants in this group received localized cold therapy using ice massage applied to the suprapubic and inner thigh regions for 20 minutes per session, three times per week for four weeks.
  Interventions: Other: Cold Stimulation
- Paraspinal Stimulation (Experimental): Participants in this group received surface electrical stimulation over the T12-L2 paraspinal region. Sessions were 30 minutes each, delivered three times per week for four weeks.
  Interventions: Other: Paraspinal Electrical Stimulation

INTERVENTIONS:
Other: Cold Stimulation — Ice massage using circular movements over the suprapubic and inner thigh areas to stimulate sensory afferents. Each session lasted 20 minutes, delivered 3 times per week for 4 weeks.
  Arms: Cold Stimulation
Other: Paraspinal Electrical Stimulation — Surface electrodes applied bilaterally to the T12-L2 region. Parameters: 20 Hz frequency, 200 µs pulse width, intensity set below motor threshold. Sessions were administered 3 times per week for 4 weeks.
  Arms: Paraspinal Stimulation

SUMMARY:
This study is being conducted to compare the effects of two simple treatments-cold therapy and electrical stimulation applied to the lower back-on sexual function and urinary control in men with spinal cord injury (SCI). Many individuals with SCI experience difficulties with erection and urinary leakage, which can negatively affect their quality of life.

In this study, participants will be assigned to receive either cold stimulation (using ice massage) or electrical stimulation over the spine. Each treatment will be applied three times a week for four weeks. The study will measure improvements in erectile function using a questionnaire called SHIM (Sexual Health Inventory for Men), and urinary control using a short-form urinary incontinence questionnaire.

The goal is to identify which treatment provides better results, is more comfortable for patients, and can be safely used as part of rehabilitation in clinical settings.

DETAILED DESCRIPTION:
Erectile dysfunction and urinary incontinence are among the most challenging secondary complications faced by men with spinal cord injury (SCI). These dysfunctions result primarily from disruption of spinal autonomic pathways and contribute significantly to reduced quality of life, social participation, and psychological well-being. Despite their clinical significance, non-invasive therapeutic approaches targeting autonomic recovery are under-researched.

This randomized controlled trial investigates the comparative effects of two non-invasive stimulation techniques-localized cold stimulation and paraspinal electrical stimulation-on erectile function and urinary incontinence in adult males with chronic SCI. Cold therapy activates superficial sensory afferents and spinal reflex arcs, while paraspinal stimulation is hypothesized to engage deeper segmental pathways within the thoracolumbar cord that contribute to pelvic organ regulation.

The study is designed to assess changes in erectile function using the SHIM questionnaire and changes in urinary incontinence using the ICIQ-UI SF. Both interventions will be applied over four weeks, with standardized protocols and session frequency. Findings from this trial may offer insight into accessible, low-risk options for addressing autonomic dysfunction in SCI and guide future rehabilitation protocols focused on quality-of-life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 25 to 55 years
* Confirmed diagnosis of thoracic or lumbar spinal cord injury (≥ 6 months post-injury)
* Presence of erectile dysfunction, indicated by a SHIM score ≤ 21
* Self-reported urinary incontinence
* Medically stable and able to participate in the study sessions

Exclusion Criteria:

* Cognitive impairment or psychiatric conditions interfering with study compliance
* Active urinary tract infection
* History of urological surgery within the past 12 months
* Presence of implanted electrical devices (e.g., pacemakers)
* Skin conditions (e.g., ulcers, dermatitis) at stimulation or ice application sites
* Use of medications affecting sexual or urinary function within the past 3 months

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Erectile Function | Baseline and after 4 weeks of intervention
  Erectile function will be assessed using the Sexual Health Inventory for Men (SHIM), a validated 5-item questionnaire measuring severity of erectile dysfunction. Scores range from 1 to 25, with higher scores indicating better function.

SECONDARY OUTCOMES:
Urinary Incontinence Severity | Baseline and after 4 weeks of intervention
  Urinary incontinence will be assessed using the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF), a validated patient-reported tool that evaluates frequency, volume of leakage, and its impact on daily life. Scores range from 0 to 21, with higher scores indicating more severe incontinence.

IPD SHARING:
Plan to Share IPD: Undecided
At this time, a definitive plan for sharing individual participant data (IPD) has not been established. Data sharing will depend on institutional policies, participant consent provisions, and ethical approval. The research team is considering options for de-identified data sharing in the future, but no repository or framework has been finalized.